CLINICAL TRIAL: NCT06846502
Title: High Power Short Duration Radiofrequency Ablation of Atrial Fibrillation Using the QDOT MICRO™ Catheter - Q-POWER STUDY
Brief Title: High Power Short Duration Radiofrequency Ablation of Atrial Fibrillation Using the QDOT MICRO™ Catheter
Acronym: Q-POWER
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Cornelis P. Allaart, Prof. dr., Amsterdam UMC, location VUmc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL76376.029.21; IIS-566 (Other Grant/Funding Number: Biosense Webster)
Record Dates: First submitted 2025-02-20; First posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-01

CONDITIONS: Atrial Fibrillation (AF)
Keywords: Atrial Fibrillation; Pulmonary Vein Isolation; Very High Power Short Duration Ablation; Cardiac Magnetic Resonance
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Paroxysmal or persistent atrial fibrillation patients (Experimental)
  Interventions: Procedure: Pulmonary vein isolation

INTERVENTIONS:
Procedure: Pulmonary vein isolation — Compared to conventional radiofrequency (RF) ablation, which is performed with a power set of 30-40 Watt for a duration of 20-30 seconds, ablation with higher power and shorter duration (vHPSD, 90W/4sec) may result in more continuous and more durable ablation lesions with a similar safety profile, while reducing procedure duration.

SUMMARY:
Atrial fibrillation (AF) is the most common cardiac arrhythmia worldwide, characterized by rapid and disorganized atrial activation leading to an irregular heart rhythm. Pulmonary vein isolation (PVI) ablation is the gold standard for catheter ablation based therapy. However, recurrence of AF after PVI is common, often due to the inability to create durable ablation lesions surrounding the pulmonary veins (PV). Conventional radiofrequency (RF) ablation is typically performed with power set at 30-40 Watt for a duration of 20-30 seconds. Previous studies have shown that ablation with very higher power and shorter duration (vHPSD, 90W/4sec) may result in more continuous and more durable ablation lesions with a similar safety profile as compared to conventional ablation lesions. This new technique may consequently improve outcomes of RF ablation for AF. Moreover, HPSD ablation of AF may significantly reduce RF duration, which could lead to shorter anaesthesia, fluoroscopy and procedure duration.

Cardiac magnetic resonance imaging (CMR) enables studying cardiac volumes, function and atrial tissue characteristics. By applying this imaging strategy before ablation, and directly (<72 hours) and later (3 months) after ablation, transient (edema) and persistent (fibrosis) effects of RF ablation in the left atrial wall and surrounding tissues may be visualized and quantified.

The Q-POWER study aims to assess the effects of VHPSD RF ablation on 1) procedural characteristics, 2) acute and long-term ablation lesion formation and collateral tissue damage as assessed by CMR and 3) clinical outcomes in AF patients.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* AF and eligible for index PVI according to current ESC guidelines

Exclusion Criteria:

* Unwilling or unable to give written informed consent
* Prior left atrial ablation
* Other left atrial arrhythmias including atrial flutters
* Prior left atrial surgery
* Severe mitral valve regurgitation
* Contraindication for gadolinium-based contrast agents
* Contraindications for CMR (including metallic implants, cochlear implants, cardiac devices, neurostimulation systems, claustrophobia)
* Renal insufficiency (eGFR < 30 ml/min)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-06-21 (Actual); Primary Completion 2024-10-28 (Actual); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Procedure duration | Procedure
  To study the effect of VHPSD ablation on procedure duration of PVI, compared with conventional Ablation Index-guided ablation.

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC, Amsterdam, North Holland, Netherlands